CLINICAL TRIAL: NCT03956342
Title: Validation of Clinician Reported Outcome (ClinRO) Measures of Pediatric Sedation
Brief Title: ClinRO Sedation Validation
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00102030
Record Dates: First submitted 2019-04-30; First posted 2019-05-20 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-04

CONDITIONS: Pediatric Sedation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pediatric Clinicians - Group 1: Pediatric clinical care clinicians who work with patients who are sedated for diagnostic or therapeutic procedures. May included, MDs, DOs, PharmDs, Nurse Practitioners, or nurses with a BSN or higher level nursing degree.
  This cohort will complete a first round of interviews to assess measure content.
- Pediatric Clinicians - Group 2: Pediatric clinical care clinicians who work with patients who are sedated for diagnostic or therapeutic procedures. May included, MDs, DOs, PharmDs, Nurse Practitioners, or nurses with a BSN or higher level nursing degree.
  This smaller cohort will be a randomized subset of the original cohort and will complete interviews to assess changes made based on the feedback from the first cohort.

SUMMARY:
This study will conduct qualitative interviews to provide evidence for the content validity and comprehension of existing physician-reported measures of sedation levels of children receiving anesthesia to facilitate a diagnostic or surgical procedure. Information gained from this study will inform the use of the measure in studies that are part of the PTN.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the content validity and physician understanding of the Pediatric Sedation State Scale (PSSS) and the University of Michigan Sedation Scale (UMSS) via cognitive interviewing methods. Qualitative Interviewers will conduct 1 hour, phone-based cognitive interviews with clinicians to assess physicians' comprehension of items and response options on clinician reported pediatric sedation scales and clinician evaluation of the relevance of the scale to capture sedation levels.

ELIGIBILITY:
Inclusion Criteria:

1. Is a practicing clinician in a clinical care environment
2. Cares for pediatric patients >50% of their time
3. Treats or works with pediatric patients who are sedated/anesthetized for diagnostic and/or therapeutic procedures
4. Holds one of the following titles/positions

   1. Anesthesiologist
   2. Pediatric critical care physician
   3. Clinical pharmacist (PharmD)
   4. Nurse anesthetist
   5. Nurse practitioner
   6. Physician assistant
   7. Nurse (with a BSN/RN or higher)
5. Is over the age of 18 years
6. Can speak English
7. Is capable of giving informed verbal consent

Exclusion Criteria:

1. Lack of access to a telephone for interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be practicing clinicians in a clinical care environment for whom >50% of their patients are sedated/anesthetized for diagnostic and/or therapeutic procedures. Clinicians may be an anesthesiologist, pediatric critical care physician, clinical pharmacist, physician assistant, nurse anesthetist, nurse practitioner, or other nurse with a BSN or higer.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Number of providers who expressed they agreed that all medically important levels of sedation are captured by the Pediatric Sedation State Scale and University of Michigan Sedation Scale as measured by a qualitative interview | 1 hour
  A 1 hour qualitative interview will be completed and coded to assess the quality of the measures being assessed.
Number of providers who expressed they understood individual sedation levels specified on the Pediatric Sedation State Scale and University of Michigan Sedation Scale as measured by a qualitative interview | 1 hour
  A 1 hour qualitative interview will be completed and coded to assess the quality of the measures being assessed.
Number of providers who expressed they understood how to complete the Pediatric Sedation State Scale and University of Michigan Sedation Scale with provided instructions as measured by a qualitative interview | 1 hour
  A 1 hour qualitative interview will be completed and coded to assess the quality of the measures being assessed. The Pediatric Sedation State Scale requires that a physician choose a level from 1 - 5 that corresponds to the patient's sedation level. The University of Michigan Sedation Scale requires that a physician choose a sedation level from 1 - 4 that corresponds to the patient's sedation level. The scales will not be completed by clinicians and will not be scored. The content of the qualitative interview is the "measure". The scales are not the measure in this study.
Number of providers who expressed any difficulty with comprehension of any of the text contained in the Pediatric Sedation State Scale or University of Michigan Sedation Scale as measured by a qualitative interview | 1 hour
  A 1 hour qualitative interview will be completed and coded to assess the quality of the measures being assessed. The Pediatric Sedation State Scale requires that a physician choose a level from 1 - 5 that corresponds to the patient's sedation level. The University of Michigan Sedation Scale requires that a physician choose a sedation level from 1 - 4 that corresponds to the patient's sedation level. The scales will not be completed by clinicians and will not be scored. The content of the qualitative interview is the "measure". The scales are not the measure in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Zigler, PhD, Principal Investigator — Duke University; Bryce B Reeve, PhD, Principal Investigator — Duke University
Locations (1):
- Imperial Building, Duke School of Medicine, Department of Population Health Sciences Office Space, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared outside of the study team.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/42/NCT03956342/Prot_SAP_000.pdf